CLINICAL TRIAL: NCT01629355
Title: Auditory Brainstem Response as a Diagnostic Tool in Schizophrenia and Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: SensoDetect (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011/2149 (REK)
Record Dates: First submitted 2012-06-06; First posted 2012-06-27 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Bipolar Disorder; Schizophrenia; Attention Deficit Disorder With Hyperactivity
Keywords: Auditory Brainstem Response; ABR; SD-BERA
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Schizophrenia: Five patients with diagnosed schizophrenia will be used to map changes in ABR/SD-BERA potentials compared to controls to establish the disease-specific pattern. Twelve patients with schizophrenia will then be studied blindly to evaluate the predictive value of the test.
- ADHD: Five patients with diagnosed ADHD will be used to map changes in ABR/SD-BERA potentials compared to controls to establish the disease-specific pattern.
- Bipolar disorder: Five patients with diagnosed Bipolar disorder will be used to map changes in ABR/SD-BERA potentials compared to controls to establish the disease-specific pattern. Twelve patients with Bipolar disorder will then be studied blindly to evaluate the predictive value of the test.
- Healthy controls: Fifteen healthy controls will be used to define normal pattern of ABR/SD-BERA potentials. Another twelve normal controls will be studied blindly to evaluate the predictive value of the test.

SUMMARY:
The purpose of this study is to study the predictive value of SensoDetect-BERA as a diagnostic tool in clinical practice for schizophrenia and bipolar disorder.

DETAILED DESCRIPTION:
Background:

Within the daily clinical work of all medical specialties, objective diagnostic tools are paramount. However, in the psychiatric field such measures are lacking. Since 1983 the method of psychoacoustics has been under development in hope to serve this purpose. A recent development of auditory brainstem response (ABR/SD-BERA), has been proposed as a potential diagnostic tool within psychiatry.

The ABR is a diagnostic tool used primarily to diagnose sensorineural hearing loss. It detects evoked potentials, generated by neuronal activity in the auditory pathways in the brainstem, within the first 10 ms following acoustic stimulation. The potentials are recorded by surface electrodes placed on the forehead and on the mastoid processes. The wave pattern recorded consists of seven peaks, which are interpreted with respect to latencies and amplitudes.

Previous studies have aimed to associate the peaks with specific anatomical structures. The method SD-BERA is a further development of the standard ABR. It uses a wider array of acoustic stimuli, including complex sounds, for instance masking noises. The measuring procedure will roughly take 25 minutes. Previous studies using these complex sounds to compare mentally healthy subjects with patients suffering from schizophrenia, ADHD and bipolar disorder have shown that the different psychiatric groups exhibit specific wave patterns.

Aims

The aim of the first study is to validate previous results and identify five (n=5) patients with diagnosed ADHD, schizophrenia and bipolar disorder, and to compare these patients (n=15) with healthy, age-matched controls.

The aim of the second study is to present a blinded study where 12 patients with schizophrenia and 12 patients with bipolar disorder (total n=24) are compared to each other and to healthy controls (n=12) in order to evaluate the method as a diagnostic tool in clinical healthcare practice.

ELIGIBILITY:
Inclusion Criteria:

* Best-practise diagnosed schizophrenia, bipolar disorder or ADHD
* Diagnosed since at least one year prior to enrollment.

Exclusion Criteria:

* Serious hearing loss
* Severe ongoing alcohol abuse or drug abuse
* Diagnosed psychiatric comorbidity
* Brain injury following cranial trauma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the University Hospital of North Norway and the General Practice Clinic in Balsfjord, Troms, Norway. Healthy controls from North Norway.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
SD-BERA patterns identified by SensoDetect using specific software | Brainstem potential patterns following an array of acoustic stimuli during a 25 min. examination
  The Auditory Brainstem Response examination (SD-BERA) will be conducted once for each patient following his/her inclusion in the study

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Wynn, M.D., Ph.D., Principal Investigator — University Hospital of North Norway
Locations (2):
- Norway (2):
  - Balsfjord Legekontor, Balsfjord, Troms
  - University Hospital North Norway, Tromsø, Troms

REFERENCES:
- [Derived] Wahlstrom V, Ahlander F, Wynn R. Auditory brainstem response as a diagnostic tool for patients suffering from schizophrenia, attention deficit hyperactivity disorder, and bipolar disorder: protocol. JMIR Res Protoc. 2015 Feb 12;4(1):e16. doi: 10.2196/resprot.3880. PMID 25679914
- See also: Abnormal auditory forward masking pattern in the brainstem response of individuals with Asperger syndrome — http://www.ncbi.nlm.nih.gov/pubmed/20628629
- See also: The Role of Psychoacoustics for the Research on Neuropsychiatric states — http://www.ncbi.nlm.nih.gov/pubmed/15146664
- See also: Aberrant brain stem functioning in schizophrenia — http://www.ncbi.nlm.nih.gov/pubmed/12467951